CLINICAL TRIAL: NCT01640197
Title: The Effects of Chronic Trans- Resveratrol Supplementation on Aspects of Cognitive Performance, Mood, Sleep, Health and Cerebral Blood Flow in Healthy, Young Humans.
Brief Title: Chronic Resveratrol Supplementation in Healthy Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Biotivia Longevity Bioceuticals (Unknown)
Responsible Party: Principal Investigator, David Kennedy, Professor, Northumbria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 22P4
Record Dates: First submitted 2012-07-10; First posted 2012-07-13 (Estimated); Results first posted 2012-10-12 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2012-08

CONDITIONS: Healthy
Keywords: Cognitive performance; Cerebral blood flow; Subjective sleep; Subjective mood; Subjective health
MeSH Terms: interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator): Methyl Cellulose administered in identical capsules as the active.
  Interventions: Other: Placebo
- 500mg resveratrol (Active Comparator): Transmax from biotivia. 500mg resveratrol (98% purity) with 10mg piperine per capsule. 1 capsule taken daily.
  Interventions: Dietary Supplement: Resveratrol

INTERVENTIONS:
Dietary Supplement: Resveratrol — Transmax (Biotivia). 500mg (1 capsule) per day for 28 days.
  Arms: 500mg resveratrol
Other: Placebo — Methyl Cellulose. 1 capsule taken once daily for 28 days.
  Arms: Placebo

SUMMARY:
The effects of chronic resveratrol supplementation have yet to be investigated in healthy humans. It is hypothesised that the effects will be different to those seen in acute supplementation. This study will look specifically at cognitive performance, cerebral blood flow, subjective sleep, mood and health, blood pressure and plasma levels of resveratrol. It is hypothesized that these measures will be affected differently by acute and chronic supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Between 18-35
* At least enrolled on undergraduate degree programme
* Native English speaker

Exclusion Criteria:

* Smoking
* Taking other medication/ supplements
* Pregnant/ breast feeding
* High caffeine consumers
* Migraine sufferers

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David O Kennedy, Professor, Principal Investigator — Northumbria University
Locations (1):
- Brain performance and nutrition research centre, Northumbria university, Newcastle upon Tyne, Tyne and Wear, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited opportunistically from Northumbria University via spam email and posters around campus.
Pre-assignment Details: Before participants were enrolled they were required to complete a training/screening session. If they met the study exclusion criteria or did not perform within the cognitive task norms (compiled from previous studies) then they were not eligible to take part in the study.
Groups:
- 500mg Resveratrol: Transmax from biotivia. 500mg resveratrol (98% purity) with 10mg piperine per capsule. 1 capsule taken daily.
  Resveratrol : Transmax (Biotivia). 500mg (1 capsule) per day for 28 days.
- Placebo: Methyl Cellulose administered in identical capsules as the active.
  Placebo : Methyl Cellulose. 1 capsule taken once daily for 28 days.
Period: Overall Study
Arm/Group | 500mg Resveratrol | Placebo
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 500mg Resveratrol | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 21.04 (2.01) | 20.00 (2.32) | 20.52 (2.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 24 | 51
  Male | 3 | 6 | 9
Region of Enrollment [Number; unit: participants]
  United Kingdom | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Chronic Modulation of Cerebral Blood Flow
Description: Cerebral blood flow (CBF) was measured in the frontal cortex with Near-Infrared Spectroscopy (NIRS). Modulation was deemed to have taken place if levels differed significantly from day 1 to day 28.
Time Frame: 40- 80 minutes post- dose on day 28 of supplementation
Population: Participants were included in the analysis if they provided full NIRS readings on session 1 and session 2.
Measure: Number; unit: Participants
Arm/Group | 500mg Resveratrol | Placebo
Number analyzed (Participants) | 22 | 24
Participants | 0 | 0
Statistical Analysis 1: Comparison: 500mg Resveratrol vs Placebo; Test type: Superiority or Other; p > 0.05, ANOVA

2. Secondary Outcome: Number of Participants With Modulated Mood
Description: Subjective mood was assessed with the Profile of mood states (POMS) questionnaire every 7 days during the 28- day period. Participants were deemed to have significant modulation of mood if their scores on week 1, week 2, week 3 and/or week 4 differed significantly from scores on the baseline questionnaire completed on day 1.
Time Frame: 28 days
Population: Participants were included in the final analysis if they had completed all questionnaires correctly.
Measure: Number; unit: Participants
Arm/Group | 500mg Resveratrol | Placebo
Number analyzed (Participants) | 26 | 28
Participants | 0 | 0
Statistical Analysis 1: Comparison: 500mg Resveratrol vs Placebo; Test type: Superiority or Other; p > 0.05, ANOVA

3. Secondary Outcome: Number of Participants With Modulated Cognitive Performance
Description: Cognitive performance was assessed by a range of cognitively demanding tasks on day 28 of the supplementation period. Participants were deemed to have significant modulation of cognitive performance if their scores on these tasks were significantly different from scores taken on day 1.
Time Frame: 28 days
Population: All participants who properly completed all repetitions of all tasks on both days were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | 500mg Resveratrol | Placebo
Number analyzed (Participants) | 22 | 19
Participants | 0 | 0
Statistical Analysis 1: Comparison: 500mg Resveratrol vs Placebo; Test type: Superiority or Other; p > 0.05, ANOVA

4. Secondary Outcome: Number of Participants With Significant Modulation of Sleep
Description: Subjective perception of sleep quality was assessed with the PSQI. Participants were deemed to have significant modulation of sleep if scores on Week 1, Week 2, Week 3 and/or Week 4 differed significantly from those on day 1 (baseline).
Time Frame: Day 28
Population: All participants who completed their questionnaires correctly were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | 500mg Resveratrol | Placebo
Number analyzed (Participants) | 25 | 28
Participants | 0 | 0
Statistical Analysis 1: Comparison: 500mg Resveratrol vs Placebo; Test type: Superiority or Other; p > 0.05, ANOVA

5. Secondary Outcome: Number of Participants With Significant Modulation of Health
Description: Subjective perceptions of health were assessed with the General Health Questionnaire. Participants were deemed to have significant modulation of health if scores on Week 1, Week 2, Week 3 and/or Week 4 differed significantly from day 1 (baseline) completion.
Time Frame: Day 28
Population: Participants were included in the analysis if they had completed questionnaires correctly.
Measure: Number; unit: Participants
Arm/Group | 500mg Resveratrol | Placebo
Number analyzed (Participants) | 25 | 28
Participants | 0 | 0
Statistical Analysis 1: Comparison: 500mg Resveratrol vs Placebo; Test type: Superiority or Other; p > 0.05, ANOVA

6. Secondary Outcome: Number of Participants With Significant Modulation of Blood Pressure
Description: Participants were deemed to have significant modulation of blood pressure if their readings on day 28 differed significantly from that taken on day 1 (baseline).
Time Frame: 28 days
Population: All participants who provided all BP readings across the study were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | 500mg Resveratrol | Placebo
Number analyzed (Participants) | 9 | 15
Participants | 0 | 0
Statistical Analysis 1: Comparison: 500mg Resveratrol vs Placebo; Test type: Superiority or Other; p > 0.05, ANOVA

7. Secondary Outcome: Number of Participants With Significant Modulation of CBF in MCA
Description: CBF was assessed in the middle cerebral artery (MCA) with Trans-cranial doppler via a trans- temporal acoustic window. Participants were deemed to have significant modulation of CBF in the MCA if readings differed significantly from those obtained on day 1 (baseline).
Time Frame: 28 days
Population: All participants who were part of the TCD component, who could provide a consistent blood flow trace, were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | 500mg Resveratrol | Placebo
Number analyzed (Participants) | 25 | 21
Participants | 0 | 0
Statistical Analysis 1: Comparison: 500mg Resveratrol vs Placebo; Test type: Superiority or Other; p > 0.05, ANOVA

ADVERSE EVENTS:
Arm/Group | 500mg Resveratrol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No